CLINICAL TRIAL: NCT00683748
Title: Monitoring Cellular Immunity After Kidney and Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Lars Wennberg, Associate Professor, Karolinska University Hospital, Department of Transplantation Surgery
Other Study IDs: T cell study
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Terminal Kidney Failure; Terminal Liver Failure
Keywords: Transplantation; Immunological monitoring; Immunological risk; T cell reactivity; Cellular immunity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Kidney transplant
- Liver transplant

SUMMARY:
After transplantation, if insufficient immunosuppression is achieved, rejection and graft loss follows. If to much immunosuppression is given, the patient suffers risk for infections and malignancies. Despite careful dosing and monitoring of drug levels, the biological effects of the immunosuppression given is difficult to predict and varies significantly. As a result, the degree of immunosuppression (or immunosuppressive status) remains unknown and clinical problems related to under- or over-immunosuppression are common. Thus, a method to determine the degree of immunosuppression would be of great and direct clinical importance and the results would be improved. T cells are the principal cells of the immunesystem causing rejection. Furthermore, all immunosuppressive regimes targets T cells. Thus, T cell reactivity could reflect the biological effects of the immunosuppression and the immunosuppressive status. In addition, T cells are of crucial importance in the immunedefence against viral diseases. Therefore, data on virus specific T cell reactivity could aid in diagnosis, monitoring and treatment of viral disease. The proposed study aim to develop a clinically useful method to monitor cellular immunity and the degree of immunosuppression after transplantation by determinations of the specific T cell reactivity to several clinically relevant viruses.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing kidney or liver transplantation at the Karolinska University Hospital

Exclusion Criteria:

* Abscence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing kidney or liver transplantation at the Karolinska University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-03 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
T cell reactivity to viral antigens | Pre-transplantation and 2 weeks, 1, 3, 6 and 12 months after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Lars Wennberg, MD, PhD, Principal Investigator — Karolinska University Hospital; Gunnar Tyden, MD, PhD, Study Director — Karolinska University Hospital
Locations (1):
- Lars Wennberg, Stockholm, Sweden